CLINICAL TRIAL: NCT05879666
Title: Improving Health and Environmental Health Literacy of Professionals
Acronym: IHEHLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Tamarra James-Todd, Primary Investigator, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB22-1510
Record Dates: First submitted 2023-04-26; First posted 2023-05-30 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reproductive Health Professionals - EHL (Experimental): All participants will complete a pre-course survey, engage in the online educational intervention, then complete 2 post-course surveys. They have the option to provide urine samples before and after the intervention.
  Interventions: Behavioral: Online educational phthalate course

INTERVENTIONS:
Behavioral: Online educational phthalate course — This is an online course focused on phthalates for reproductive health professionals. It consists of videos from patient, scientist, and OBGYN perspectives describing how phthalates relate to reproductive health. There is also an interactive module and worksheet to facilitate conversations about phthalates with pregnant individuals.

SUMMARY:
The goal of this clinical trial is to understand the impact of an educational intervention on reproductive health care providers' environmental health literacy related to phthalates. The main questions to answer are:

1. Does a web-based educational intervention improve the environmental health literacy of personal care product chemicals based on pre/post/post intervention survey data?
2. Does a web-based educational intervention improve reproductive health professionals' confidence and awareness for communication to patients on environmental health literacy?
3. Do concentrations of personal care product chemicals in reproductive health professionals decrease after the web-based educational intervention?

Participants will be asked to complete three surveys: one before the educational intervention, and two after the intervention. The will be asked to complete the approximately 1-hour online educational intervention, which consists of a series of videos from the perspectives of patients, OBGYNs, and researchers, an interactive module, and a worksheet to facilitate conversation with patients.

ELIGIBILITY:
Inclusion Criteria:

* Employed in a patient-facing role relevant to reproductive health care (e.g., obstetricians, gynecologists, medical assistants, doulas, and nurses, etc.)

Exclusion Criteria:

* Practitioner does not interact with patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Baseline phthalate environmental health literacy | Up to 2 weeks
  Measure of phthalate reproductive environmental health literacy via validated scale (pre educational intervention), the Phthalate Environmental Reproductive Health Literacy (PERHL) scale. Scores on the PERHL scale range from 6-31, with a higher score indicating higher environmental health literacy.
Change from baseline phthalate environmental health literacy | Up to 4 weeks
  Measure of phthalate reproductive environmental health literacy via validated scale (post educational intervention), the Phthalate Environmental Reproductive Health Literacy (PERHL) scale. Scores on the PERHL scale range from 6-31, with a higher score indicating higher environmental health literacy.
Sustained change from baseline phthalate environmental health literacy | 2 months
  Measure of phthalate reproductive environmental health literacy via validated scale (2 months post educational intervention), the Phthalate Environmental Reproductive Health Literacy (PERHL) scale. Scores on the PERHL scale range from 6-31, with a higher score indicating higher environmental health literacy.
Baseline urinary biomarkers of phthalate exposure | Up to 2 weeks
  Collected via urine samples, measure of previous phthalate exposures. We will evaluate urine samples for urinary phthalate metabolite concentrations using a standard panel, measuring 16 urinary phthalate metabolites and their replacements (CX-MINCH, MECPTP, MEHHTP, OH-MINCH, mBP, mBzP, mCnP, mCOP, mCPP, mECPP, mEHHP, mEHP, mEOHP, mEP, mNP, miBP), and assayed using a modified method from the Centers for Disease Control and Prevention. Briefly, HPLC-MS/MS ESI is conducted based on the CDC's Phthalate Metabolites in Urine Method No: 6306.03. We will also calculate the molar sums of SG-adjusted metabolites representing metabolites related to parent compound DEHP (i.e., ΣDEHP = (mEHP/278) + (mEHHP/294) + (mEOHP/292) + (mECPP/308)) and personal care product (PCP)-associated phthalates (i.e., ΣPCP = (mBP/222) + (miBP/222) + (mEP/194)). Units for all metabolites will be ng/mL.
Change in urinary biomarkers of phthalate exposure | Up to 4 weeks
  Collected via urine samples, measure of previous phthalate exposures. We will evaluate urine samples for urinary phthalate metabolite concentrations using a standard panel, measuring 16 urinary phthalate metabolites and their replacements (CX-MINCH, MECPTP, MEHHTP, OH-MINCH, mBP, mBzP, mCnP, mCOP, mCPP, mECPP, mEHHP, mEHP, mEOHP, mEP, mNP, miBP), and assayed using a modified method from the Centers for Disease Control and Prevention. Briefly, HPLC-MS/MS ESI is conducted based on the CDC's Phthalate Metabolites in Urine Method No: 6306.03. We will also calculate the molar sums of SG-adjusted metabolites representing metabolites related to parent compound DEHP (i.e., ΣDEHP = (mEHP/278) + (mEHHP/294) + (mEOHP/292) + (mECPP/308)) and personal care product (PCP)-associated phthalates (i.e., ΣPCP = (mBP/222) + (miBP/222) + (mEP/194)). Units for all metabolites will be ng/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard T.H. Chan School of Public Health, Boston, Massachusetts, United States